CLINICAL TRIAL: NCT00033085
Title: Double-Blind, Placebo-Controlled Trial of Ondansetron for the Treatment of Cocaine Dependence
Brief Title: Ondansetron for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0005-1; NCT00024726 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Cocaine-Related Disorders; Drug Administration Schedule
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ondansetron

INTERVENTIONS:
Drug: Ondansetron

SUMMARY:
The purpose of this study is to assess the efficacy and safety of ondansetron to reduce cocaine use in subjects with cocaine dependence.

DETAILED DESCRIPTION:
Double-blind, placebo-controlled, 4-parallel group design to assess the efficacy and safety of 3 wide range doses of ondansetron to reduce cocaine use in subjects with cocaine dependence and to determine the optimal dose of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

Male/Female, at least 18 yrs of age; DSM-4 diagnosis of cocaine dependence; seeking Treatment for cocaine dependence; have ability to understand, having understood and provide written consent; females of child bearing potential that use accepted method of birth control

Exclusion Criteria:

Additional criteria available during screening at the site.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-05; Study Completion 2002-12

PRIMARY OUTCOMES:
Cocaine use

CONTACTS AND LOCATIONS:
Overall Officials: John Roache, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Hlth Sci Ctr San Ant, San Antonio, Texas, United States